CLINICAL TRIAL: NCT02131259
Title: Post Marketing Surveillance on Long Term Drug Use of GIOTRIF Tablets in Patients With Epidermal Growth Factor Receptor Mutation-positive Inoperable or Recurrent Non-small Cell Lung Cancer.
Brief Title: Long-term Observation PMS for Afatinib
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200.181
Record Dates: First submitted 2014-05-05; First posted 2014-05-06 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Afatinib
  Interventions: Drug: Afatinib dimaleate

INTERVENTIONS:
Drug: Afatinib dimaleate — 20mg - 50mg

SUMMARY:
In Japan, post-approval execution of post marketing surveillance (PMS) is requested by the Japanese Pharmaceutical Affairs Law (J-PAL) in order to accumulate safety and efficacy data for reexamination. Reexamination period is defined by J-PAL. Eight years after approval of a new substance, results of PMS need to be submitted as a part of reexamination dossier to the Japanese regulatory authority, the Ministry of Health, Labour and Welfare (MHLW).

ELIGIBILITY:
Inclusion criteria:

- Patients with Epidermal Growth Factor Receptor (EGFR) mutation-positive inoperable or recurrent non-small cell lung cancer (NSCLC)will be included.

Exclusion criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1500
Sampling Method: Non-Probability Sample
Enrollment: 1605 (Actual)
Dates: Start 2014-05-07 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (432):
- Japan (432):
  - Boehringer Ingelheim Investigational Site 145, Adachi Tokyo
  - Boehringer Ingelheim Investigational Site 429, Aira Kagoshima
  - Boehringer Ingelheim Investigational Site 64, Aizuwakamatsu Fukushima
  - Boehringer Ingelheim Investigational Site 44, Akita Akita
  - Boehringer Ingelheim Investigational Site 45, Akita Akita
  - Boehringer Ingelheim Investigational Site 46, Akita Akita
  - Boehringer Ingelheim Investigational Site 47, Akita Akita
  - Boehringer Ingelheim Investigational Site 333, Amagasaki Hyogo
  - Boehringer Ingelheim Investigational Site 266, Anjo Aichi
  - Boehringer Ingelheim Investigational Site 27, Aomori Aomori
  - Boehringer Ingelheim Investigational Site 28, Aomori Aomori
  - Boehringer Ingelheim Investigational Site 127, Asahi Chiba
  - Boehringer Ingelheim Investigational Site 128, Asahi Chiba
  - Boehringer Ingelheim Investigational Site 18, Asahikawa Hokkaido
  - Boehringer Ingelheim Investigational Site 19, Asahikawa Hokkaido
  - Boehringer Ingelheim Investigational Site 20, Asahikawa Hokkaido
  - Boehringer Ingelheim Investigational Site 21, Asahikawa Hokkaido
  - Boehringer Ingelheim Investigational Site 198, Atsugi Kanagawa
  - Boehringer Ingelheim Investigational Site 294, Ayabe Kyoto
  - Boehringer Ingelheim Investigational Site 142, Bunkyo Tokyo
  - Boehringer Ingelheim Investigational Site 143, Bunkyo Tokyo
  - Boehringer Ingelheim Investigational Site 144, Bunkyo Tokyo
  - Boehringer Ingelheim Investigational Site 112, Chiba Chiba
  - Boehringer Ingelheim Investigational Site 113, Chiba Chiba
  - Boehringer Ingelheim Investigational Site 114, Chiba Chiba
  - Boehringer Ingelheim Investigational Site 115, Chiba Chiba
  - Boehringer Ingelheim Investigational Site 116, Chiba Chiba
  - Boehringer Ingelheim Investigational Site 117, Chiba Chiba
  - Boehringer Ingelheim Investigational Site 402, Chikugo Fukuoka
  - Boehringer Ingelheim Investigational Site 16, Chitose Hokkaido
  - Boehringer Ingelheim Investigational Site 132, Chiyoda Tokyo
  - Boehringer Ingelheim Investigational Site 133, Chiyoda Tokyo
  - Boehringer Ingelheim Investigational Site 134, Chiyoda Tokyo
  - Boehringer Ingelheim Investigational Site 135, Chuo Tokyo
  - Boehringer Ingelheim Investigational Site 136, Chuo Tokyo
  - Boehringer Ingelheim Investigational Site 234, Chuo Yamanashi
  - Boehringer Ingelheim Investigational Site 235, Chuo Yamanashi
  - Boehringer Ingelheim Investigational Site 48, Daisen Akita
  - Boehringer Ingelheim Investigational Site 147, Edogawa Tokyo
  - Boehringer Ingelheim Investigational Site 148, Edogawa Tokyo
  - Boehringer Ingelheim Investigational Site 173, Fuchu Tokyo
  - Boehringer Ingelheim Investigational Site 257, Fuji Shizuoka
  - Boehringer Ingelheim Investigational Site 260, Fujieda Shizuoka
  - Boehringer Ingelheim Investigational Site 97, Fujioka Gumma
  - Boehringer Ingelheim Investigational Site 203, Fujisawa Kanagawa
  - Boehringer Ingelheim Investigational Site 111, Fukaya Saitama
  - Boehringer Ingelheim Investigational Site 231, Fukui Fukui
  - Boehringer Ingelheim Investigational Site 232, Fukui Fukui
  - Boehringer Ingelheim Investigational Site 393, Fukuoka Fukuoka
  - Boehringer Ingelheim Investigational Site 394, Fukuoka Fukuoka
  - Boehringer Ingelheim Investigational Site 395, Fukuoka Fukuoka
  - Boehringer Ingelheim Investigational Site 396, Fukuoka Fukuoka
  - Boehringer Ingelheim Investigational Site 399, Fukuoka Fukuoka
  - Boehringer Ingelheim Investigational Site 58, Fukushima Fukushima
  - Boehringer Ingelheim Investigational Site 59, Fukushima Fukushima
  - Boehringer Ingelheim Investigational Site 60, Fukushima Fukushima
  - Boehringer Ingelheim Investigational Site 356, Fukuyama Hiroshima
  - Boehringer Ingelheim Investigational Site 357, Fukuyama Hiroshima
  - Boehringer Ingelheim Investigational Site 121, Funabashi Chiba
  - Boehringer Ingelheim Investigational Site 251, Gifu Gifu
  - Boehringer Ingelheim Investigational Site 252, Gifu Gifu
  - Boehringer Ingelheim Investigational Site 432, Ginowan Okinawa
  - Boehringer Ingelheim Investigational Site 321, Habikino Osaka
  - Boehringer Ingelheim Investigational Site 29, Hachinohe Aomori
  - Boehringer Ingelheim Investigational Site 30, Hachinohe Aomori
  - Boehringer Ingelheim Investigational Site 176, Hachioji Tokyo
  - Boehringer Ingelheim Investigational Site 209, Hadano Kanagawa
  - Boehringer Ingelheim Investigational Site 3, Hakodate Hokkaido
  - Boehringer Ingelheim Investigational Site 349, Hamada Shimane
  - Boehringer Ingelheim Investigational Site 261, Hamamatsu Shizuoka
  - Boehringer Ingelheim Investigational Site 367, Hatsukaichi Hiroshima
  - Boehringer Ingelheim Investigational Site 107, Hidaka Saitama
  - Boehringer Ingelheim Investigational Site 76, Higashiibaraki Ibaraki
  - Boehringer Ingelheim Investigational Site 53, Higashiokitama Yamagata
  - Boehringer Ingelheim Investigational Site 54, Higashiokitama Yamagata
  - Boehringer Ingelheim Investigational Site 318, Higashiosaka Osaka
  - Boehringer Ingelheim Investigational Site 339, Himeji Hyogo
  - Boehringer Ingelheim Investigational Site 316, Hirakata Osaka
  - Boehringer Ingelheim Investigational Site 317, Hirakata Osaka
  - Boehringer Ingelheim Investigational Site 208, Hiratsuka Kanagawa
  - Boehringer Ingelheim Investigational Site 31, Hirosaki Aomori
  - Boehringer Ingelheim Investigational Site 32, Hirosaki Aomori
  - Boehringer Ingelheim Investigational Site 359, Hiroshima Hiroshima
  - Boehringer Ingelheim Investigational Site 360, Hiroshima Hiroshima
  - Boehringer Ingelheim Investigational Site 361, Hiroshima Hiroshima
  - Boehringer Ingelheim Investigational Site 362, Hiroshima Hiroshima
  - Boehringer Ingelheim Investigational Site 363, Hiroshima Hiroshima
  - Boehringer Ingelheim Investigational Site 364, Hiroshima Hiroshima
  - Boehringer Ingelheim Investigational Site 79, Hitachi Ibaraki
  - Boehringer Ingelheim Investigational Site 77, Hitachinaka Ibaraki
  - Boehringer Ingelheim Investigational Site 78, Hitachinaka Ibaraki
  - Boehringer Ingelheim Investigational Site 312, Ibaraki Osaka
  - Boehringer Ingelheim Investigational Site 131, Ichihara Chiba
  - Boehringer Ingelheim Investigational Site 120, Ichikawa Chiba
  - Boehringer Ingelheim Investigational Site 246, Iida Nagano
  - Boehringer Ingelheim Investigational Site 247, Iida Nagano
  - Boehringer Ingelheim Investigational Site 309, Ikeda Osaka
  - Boehringer Ingelheim Investigational Site 248, Ina Nagano
  - Boehringer Ingelheim Investigational Site 118, Inzai Chiba
  - Boehringer Ingelheim Investigational Site 105, Iruma Saitama
  - Boehringer Ingelheim Investigational Site 428, Isa Kagoshima
  - Boehringer Ingelheim Investigational Site 407, Isahaya Nagasaki
  - Boehringer Ingelheim Investigational Site 281, Ise Mie
  - Boehringer Ingelheim Investigational Site 95, Isesaki Gumma
  - Boehringer Ingelheim Investigational Site 168, Itabashi Tokyo
  - Boehringer Ingelheim Investigational Site 65, Iwaki Fukushima
  - Boehringer Ingelheim Investigational Site 368, Iwakuni Yamaguchi
  - Boehringer Ingelheim Investigational Site 17, Iwamizawa Hokkaido
  - Boehringer Ingelheim Investigational Site 324, Izumi Osaka
  - Boehringer Ingelheim Investigational Site 348, Izumo Shimane
  - Boehringer Ingelheim Investigational Site 255, Izunokuni Shizuoka
  - Boehringer Ingelheim Investigational Site 213, Joetsu Niigata
  - Boehringer Ingelheim Investigational Site 214, Joetsu Niigata
  - Boehringer Ingelheim Investigational Site 289, Joyo Kyoto
  - Boehringer Ingelheim Investigational Site 422, Kagoshima Kagoshima
  - Boehringer Ingelheim Investigational Site 423, Kagoshima Kagoshima
  - Boehringer Ingelheim Investigational Site 424, Kagoshima Kagoshima
  - Boehringer Ingelheim Investigational Site 425, Kagoshima Kagoshima
  - Boehringer Ingelheim Investigational Site 426, Kagoshima Kagoshima
  - Boehringer Ingelheim Investigational Site 262, Kakegawa Shizuoka
  - Boehringer Ingelheim Investigational Site 340, Kakogawa Hyogo
  - Boehringer Ingelheim Investigational Site 201, Kamakura Kanagawa
  - Boehringer Ingelheim Investigational Site 202, Kamakura Kanagawa
  - Boehringer Ingelheim Investigational Site 130, Kamogawa Chiba
  - Boehringer Ingelheim Investigational Site 223, Kanazawa Ishikawa
  - Boehringer Ingelheim Investigational Site 224, Kanazawa Ishikawa
  - Boehringer Ingelheim Investigational Site 225, Kanazawa Ishikawa
  - Boehringer Ingelheim Investigational Site 226, Kanazawa Ishikawa
  - Boehringer Ingelheim Investigational Site 227, Kanazawa Ishikawa
  - Boehringer Ingelheim Investigational Site 74, Kasama Ibaraki
  - Boehringer Ingelheim Investigational Site 343, Kashihara Nara
  - Boehringer Ingelheim Investigational Site 123, Kashiwa Chiba
  - Boehringer Ingelheim Investigational Site 124, Kashiwa Chiba
  - Boehringer Ingelheim Investigational Site 125, Kashiwa Chiba
  - Boehringer Ingelheim Investigational Site 104, Kasukabe Saitama
  - Boehringer Ingelheim Investigational Site 106, Kawagoe Saitama
  - Boehringer Ingelheim Investigational Site 100, Kawaguchi Saitama
  - Boehringer Ingelheim Investigational Site 99, Kawaguchi Saitama
  - Boehringer Ingelheim Investigational Site 182, Kawasaki Kanagawa
  - Boehringer Ingelheim Investigational Site 183, Kawasaki Kanagawa
  - Boehringer Ingelheim Investigational Site 184, Kawasaki Kanagawa
  - Boehringer Ingelheim Investigational Site 185, Kawasaki Kanagawa
  - Boehringer Ingelheim Investigational Site 186, Kawasaki Kanagawa
  - Boehringer Ingelheim Investigational Site 42, Kesennuma Miyagi
  - Boehringer Ingelheim Investigational Site 129, Kisarazu Chiba
  - Boehringer Ingelheim Investigational Site 325, Kishiwada Osaka
  - Boehringer Ingelheim Investigational Site 326, Kishiwada Osaka
  - Boehringer Ingelheim Investigational Site 377, Kita Kagawa
  - Boehringer Ingelheim Investigational Site 110, Kitaadachi Saitama
  - Boehringer Ingelheim Investigational Site 387, Kitakyushu Fukuoka
  - Boehringer Ingelheim Investigational Site 388, Kitakyushu Fukuoka
  - Boehringer Ingelheim Investigational Site 389, Kitakyushu Fukuoka
  - Boehringer Ingelheim Investigational Site 390, Kitakyushu Fukuoka
  - Boehringer Ingelheim Investigational Site 391, Kitakyushu Fukuoka
  - Boehringer Ingelheim Investigational Site 392, Kitakyushu Fukuoka
  - Boehringer Ingelheim Investigational Site 25, Kitami Hokkaido
  - Boehringer Ingelheim Investigational Site 26, Kitami Hokkaido
  - Boehringer Ingelheim Investigational Site 180, Kiyose Tokyo
  - Boehringer Ingelheim Investigational Site 181, Kiyose Tokyo
  - Boehringer Ingelheim Investigational Site 327, Kobe Hyogo
  - Boehringer Ingelheim Investigational Site 328, Kobe Hyogo
  - Boehringer Ingelheim Investigational Site 329, Kobe Hyogo
  - Boehringer Ingelheim Investigational Site 330, Kobe Hyogo
  - Boehringer Ingelheim Investigational Site 331, Kobe Hyogo
  - Boehringer Ingelheim Investigational Site 383, Kochi Kochi
  - Boehringer Ingelheim Investigational Site 384, Kochi Kochi
  - Boehringer Ingelheim Investigational Site 385, Kochi Kochi
  - Boehringer Ingelheim Investigational Site 386, Kochi Kochi
  - Boehringer Ingelheim Investigational Site 174, Kodaira Tokyo
  - Boehringer Ingelheim Investigational Site 233, Kofu Yamanashi
  - Boehringer Ingelheim Investigational Site 397, Koga Fukuoka
  - Boehringer Ingelheim Investigational Site 398, Koga Fukuoka
  - Boehringer Ingelheim Investigational Site 179, Komae Tokyo
  - Boehringer Ingelheim Investigational Site 228, Komatsu Ishikawa
  - Boehringer Ingelheim Investigational Site 61, Koriyama Fukushima
  - Boehringer Ingelheim Investigational Site 62, Koriyama Fukushima
  - Boehringer Ingelheim Investigational Site 63, Koriyama Fukushima
  - Boehringer Ingelheim Investigational Site 103, Koshigaya Saitama
  - Boehringer Ingelheim Investigational Site 149, Koto Tokyo
  - Boehringer Ingelheim Investigational Site 150, Koto Tokyo
  - Boehringer Ingelheim Investigational Site 108, Kumagaya Saitama
  - Boehringer Ingelheim Investigational Site 109, Kumagaya Saitama
  - Boehringer Ingelheim Investigational Site 411, Kumamoto Kumamoto
  - Boehringer Ingelheim Investigational Site 413, Kumamoto Kumamoto
  - Boehringer Ingelheim Investigational Site 414, Kumamoto Kumamoto
  - Boehringer Ingelheim Investigational Site 415, Kumamoto Kumamoto
  - Boehringer Ingelheim Investigational Site 352, Kurashiki Okayama
  - Boehringer Ingelheim Investigational Site 355, Kurashiki Okayama
  - Boehringer Ingelheim Investigational Site 365, Kure Hiroshima
  - Boehringer Ingelheim Investigational Site 366, Kure Hiroshima
  - Boehringer Ingelheim Investigational Site 24, Kushiro
  - Boehringer Ingelheim Investigational Site 278, Kuwana Mie
  - Boehringer Ingelheim Investigational Site 285, Kyoto Kyoto
  - Boehringer Ingelheim Investigational Site 286, Kyoto Kyoto
  - Boehringer Ingelheim Investigational Site 287, Kyoto Kyoto
  - Boehringer Ingelheim Investigational Site 288, Kyoto Kyoto
  - Boehringer Ingelheim Investigational Site 291, Kyoto Kyoto
  - Boehringer Ingelheim Investigational Site 292, Kyoto Kyoto
  - Boehringer Ingelheim Investigational Site 293, Kyoto Kyoto
  - Boehringer Ingelheim Investigational Site 177, Machida Tokyo
  - Boehringer Ingelheim Investigational Site 91, Maebashi Gumma
  - Boehringer Ingelheim Investigational Site 92, Maebashi Gumma
  - Boehringer Ingelheim Investigational Site 93, Maebashi Gumma
  - Boehringer Ingelheim Investigational Site 94, Maebashi Gumma
  - Boehringer Ingelheim Investigational Site 119, Matsudo Chiba
  - Boehringer Ingelheim Investigational Site 346, Matsue Shimane
  - Boehringer Ingelheim Investigational Site 347, Matsue Shimane
  - Boehringer Ingelheim Investigational Site 241, Matsumoto Nagano
  - Boehringer Ingelheim Investigational Site 242, Matsumoto Nagano
  - Boehringer Ingelheim Investigational Site 243, Matsumoto Nagano
  - Boehringer Ingelheim Investigational Site 244, Matsumoto Nagano
  - Boehringer Ingelheim Investigational Site 249, Matsumoto Nagano
  - Boehringer Ingelheim Investigational Site 250, Matsumoto Nagano
  - Boehringer Ingelheim Investigational Site 280, Matsusaka Mie
  - Boehringer Ingelheim Investigational Site 378, Matsuyama Ehime
  - Boehringer Ingelheim Investigational Site 379, Matsuyama Ehime
  - Boehringer Ingelheim Investigational Site 381, Matsuyama Ehime
  - Boehringer Ingelheim Investigational Site 158, Meguro Tokyo
  - Boehringer Ingelheim Investigational Site 159, Meguro Tokyo
  - Boehringer Ingelheim Investigational Site 416, Minamata Kumamoto
  - Boehringer Ingelheim Investigational Site 137, Minato Tokyo
  - Boehringer Ingelheim Investigational Site 138, Minato Tokyo
  - Boehringer Ingelheim Investigational Site 139, Minato Tokyo
  - Boehringer Ingelheim Investigational Site 140, Minato Tokyo
  - Boehringer Ingelheim Investigational Site 171, Mitaka Tokyo
  - Boehringer Ingelheim Investigational Site 172, Mitaka Tokyo
  - Boehringer Ingelheim Investigational Site 75, Mito Ibaraki
  - Boehringer Ingelheim Investigational Site 419, Miyazaki Miyazaki
  - Boehringer Ingelheim Investigational Site 420, Miyazaki Miyazaki
  - Boehringer Ingelheim Investigational Site 421, Miyazaki Miyazaki
  - Boehringer Ingelheim Investigational Site 315, Moriguchi Osaka
  - Boehringer Ingelheim Investigational Site 33, Morioka Iwate
  - Boehringer Ingelheim Investigational Site 34, Morioka Iwate
  - Boehringer Ingelheim Investigational Site 282, Moriyama Shiga
  - Boehringer Ingelheim Investigational Site 283, Moriyama Shiga
  - Boehringer Ingelheim Investigational Site 5, Muroran Hokkaido
  - Boehringer Ingelheim Investigational Site 284, Nagahama Shiga
  - Boehringer Ingelheim Investigational Site 274, Nagakute Aichi
  - Boehringer Ingelheim Investigational Site 236, Nagano Nagano
  - Boehringer Ingelheim Investigational Site 237, Nagano Nagano
  - Boehringer Ingelheim Investigational Site 238, Nagano Nagano
  - Boehringer Ingelheim Investigational Site 210, Nagaoka Niigata
  - Boehringer Ingelheim Investigational Site 211, Nagaoka Niigata
  - Boehringer Ingelheim Investigational Site 212, Nagaoka Niigata
  - Boehringer Ingelheim Investigational Site 405, Nagasaki Nagasaki
  - Boehringer Ingelheim Investigational Site 406, Nagasaki Nagasaki
  - Boehringer Ingelheim Investigational Site 267, Nagoya Aichi
  - Boehringer Ingelheim Investigational Site 268, Nagoya Aichi
  - Boehringer Ingelheim Investigational Site 269, Nagoya Aichi
  - Boehringer Ingelheim Investigational Site 270, Nagoya Aichi
  - Boehringer Ingelheim Investigational Site 271, Nagoya Aichi
  - Boehringer Ingelheim Investigational Site 272, Nagoya Aichi
  - Boehringer Ingelheim Investigational Site 80, Naka Ibaraki
  - Boehringer Ingelheim Investigational Site 167, Nakano Tokyo
  - Boehringer Ingelheim Investigational Site 341, Nara Nara
  - Boehringer Ingelheim Investigational Site 122, Narashino Chiba
  - Boehringer Ingelheim Investigational Site 39, Natori Miyagi
  - Boehringer Ingelheim Investigational Site 169, Nerima Tokyo
  - Boehringer Ingelheim Investigational Site 170, Nerima Tokyo
  - Boehringer Ingelheim Investigational Site 215, Niigata Niigata
  - Boehringer Ingelheim Investigational Site 216, Niigata Niigata
  - Boehringer Ingelheim Investigational Site 217, Niigata Niigata
  - Boehringer Ingelheim Investigational Site 218, Niigata Niigata
  - Boehringer Ingelheim Investigational Site 382, Niihama Ehime
  - Boehringer Ingelheim Investigational Site 334, Nishinomiya Hyogo
  - Boehringer Ingelheim Investigational Site 335, Nishinomiya Hyogo
  - Boehringer Ingelheim Investigational Site 336, Nishinomiya Hyogo
  - Boehringer Ingelheim Investigational Site 22, Obihiro Hokkaido
  - Boehringer Ingelheim Investigational Site 23, Obihiro Hokkaido
  - Boehringer Ingelheim Investigational Site 253, Ogaki Gifu
  - Boehringer Ingelheim Investigational Site 417, Oita Oita
  - Boehringer Ingelheim Investigational Site 418, Oita Oita
  - Boehringer Ingelheim Investigational Site 350, Okayama Okayama
  - Boehringer Ingelheim Investigational Site 351, Okayama Okayama
  - Boehringer Ingelheim Investigational Site 353, Okayama Okayama
  - Boehringer Ingelheim Investigational Site 264, Okazaki Aichi
  - Boehringer Ingelheim Investigational Site 265, Okazaki Aichi
  - Boehringer Ingelheim Investigational Site 178, Ome Tokyo
  - Boehringer Ingelheim Investigational Site 358, Onomichi Hiroshima
  - Boehringer Ingelheim Investigational Site 295, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 296, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 297, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 298, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 299, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 300, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 301, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 302, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 303, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 304, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 305, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 306, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 307, Osaka Osaka
  - Boehringer Ingelheim Investigational Site 43, Osaki Miyagi
  - Boehringer Ingelheim Investigational Site 35, Oshu Iwate
  - Boehringer Ingelheim Investigational Site 96, Ota Gumma
  - Boehringer Ingelheim Investigational Site 153, Ota Tokyo
  - Boehringer Ingelheim Investigational Site 154, Ota Tokyo
  - Boehringer Ingelheim Investigational Site 155, Ota Tokyo
  - Boehringer Ingelheim Investigational Site 156, Ota Tokyo
  - Boehringer Ingelheim Investigational Site 4, Otaru Hokkaido
  - Boehringer Ingelheim Investigational Site 85, Otawara Tochigi
  - Boehringer Ingelheim Investigational Site 70, Ryugasaki Ibaraki
  - Boehringer Ingelheim Investigational Site 403, Saga Saga
  - Boehringer Ingelheim Investigational Site 204, Sagamihara Kanagawa
  - Boehringer Ingelheim Investigational Site 205, Sagamihara Kanagawa
  - Boehringer Ingelheim Investigational Site 206, Sagamihara Kanagawa
  - Boehringer Ingelheim Investigational Site 207, Sagamihara Kanagawa
  - Boehringer Ingelheim Investigational Site 322, Sakai Osaka
  - Boehringer Ingelheim Investigational Site 323, Sakai Osaka
  - Boehringer Ingelheim Investigational Site 56, Sakata
  - Boehringer Ingelheim Investigational Site 57, Sakata
  - Boehringer Ingelheim Investigational Site 239, Saku Nagano
  - Boehringer Ingelheim Investigational Site 126, Sakura Chiba
  - Boehringer Ingelheim Investigational Site 338, Sanda Hyogo
  - Boehringer Ingelheim Investigational Site 10, Sapporo Hokkaido
  - Boehringer Ingelheim Investigational Site 11, Sapporo Hokkaido
  - Boehringer Ingelheim Investigational Site 12, Sapporo Hokkaido
  - Boehringer Ingelheim Investigational Site 13, Sapporo Hokkaido
  - Boehringer Ingelheim Investigational Site 14, Sapporo Hokkaido
  - Boehringer Ingelheim Investigational Site 15, Sapporo Hokkaido
  - Boehringer Ingelheim Investigational Site 1, Sapporo Hokkaido
  - Boehringer Ingelheim Investigational Site 2, Sapporo Hokkaido
  - Boehringer Ingelheim Investigational Site 7, Sapporo Hokkaido
  - Boehringer Ingelheim Investigational Site 8, Sapporo Hokkaido
  - Boehringer Ingelheim Investigational Site 9, Sapporo Hokkaido
  - Boehringer Ingelheim Investigational Site 409, Sasebo Nagasaki
  - Boehringer Ingelheim Investigational Site 410, Sasebo Nagasaki
  - Boehringer Ingelheim Investigational Site 73, Sashima Ibaraki
  - Boehringer Ingelheim Investigational Site 427, Satsumasendai Kagoshima
  - Boehringer Ingelheim Investigational Site 36, Sendai Miyagi
  - Boehringer Ingelheim Investigational Site 37, Sendai Miyagi
  - Boehringer Ingelheim Investigational Site 38, Sendai Miyagi
  - Boehringer Ingelheim Investigational Site 40, Sendai Miyagi
  - Boehringer Ingelheim Investigational Site 275, Seto Aichi
  - Boehringer Ingelheim Investigational Site 219, Shibata Niigata
  - Boehringer Ingelheim Investigational Site 98, Shibukawa Gumma
  - Boehringer Ingelheim Investigational Site 157, Shibuya Tokyo
  - Boehringer Ingelheim Investigational Site 408, Shimabara Nagasaki
  - Boehringer Ingelheim Investigational Site 430, Shimajiri Okinawa
  - Boehringer Ingelheim Investigational Site 369, Shimonoseki Yamaguchi
  - Boehringer Ingelheim Investigational Site 371, Shimonoseki Yamaguchi
  - Boehringer Ingelheim Investigational Site 372, Shimonoseki Yamaguchi
  - Boehringer Ingelheim Investigational Site 83, Shimotsuga Tochigi
  - Boehringer Ingelheim Investigational Site 84, Shimotsuga Tochigi
  - Boehringer Ingelheim Investigational Site 87, Shimotsuke Tochigi
  - Boehringer Ingelheim Investigational Site 88, Shimotsuke Tochigi
  - Boehringer Ingelheim Investigational Site 151, Shinagawa Tokyo
  - Boehringer Ingelheim Investigational Site 152, Shinagawa Tokyo
  - Boehringer Ingelheim Investigational Site 160, Shinjuku Tokyo
  - Boehringer Ingelheim Investigational Site 161, Shinjuku Tokyo
  - Boehringer Ingelheim Investigational Site 162, Shinjuku Tokyo
  - Boehringer Ingelheim Investigational Site 163, Shinjuku Tokyo
  - Boehringer Ingelheim Investigational Site 164, Shinjuku Tokyo
  - Boehringer Ingelheim Investigational Site 165, Shinjuku Tokyo
  - Boehringer Ingelheim Investigational Site 166, Shinjuku Tokyo
  - Boehringer Ingelheim Investigational Site 41, Shiogama Miyagi
  - Boehringer Ingelheim Investigational Site 258, Shizuoka Shizuoka
  - Boehringer Ingelheim Investigational Site 259, Shizuoka Shizuoka
  - Boehringer Ingelheim Investigational Site 102, Soka Saitama
  - Boehringer Ingelheim Investigational Site 310, Suita Osaka
  - Boehringer Ingelheim Investigational Site 311, Suita Osaka
  - Boehringer Ingelheim Investigational Site 146, Sumida Tokyo
  - Boehringer Ingelheim Investigational Site 332, Sumoto Hyogo
  - Boehringer Ingelheim Investigational Site 256, Sunto Shizuoka
  - Boehringer Ingelheim Investigational Site 245, Suwa Nagano
  - Boehringer Ingelheim Investigational Site 175, Tachikawa Tokyo
  - Boehringer Ingelheim Investigational Site 141, Taito Tokyo
  - Boehringer Ingelheim Investigational Site 376, Takamatsu Kagawa
  - Boehringer Ingelheim Investigational Site 222, Takaoka Toyama
  - Boehringer Ingelheim Investigational Site 337, Takarazuka Hyogo
  - Boehringer Ingelheim Investigational Site 89, Takasaki Gumma
  - Boehringer Ingelheim Investigational Site 90, Takasaki Gumma
  - Boehringer Ingelheim Investigational Site 313, Takatsuki Osaka
  - Boehringer Ingelheim Investigational Site 314, Takatsuki Osaka
  - Boehringer Ingelheim Investigational Site 254, Takayama Gifu
  - Boehringer Ingelheim Investigational Site 342, Tenri Nara
  - Boehringer Ingelheim Investigational Site 86, Tochigi Tochigi
  - Boehringer Ingelheim Investigational Site 101, Toda Saitama
  - Boehringer Ingelheim Investigational Site 373, Tokushima Tokushima
  - Boehringer Ingelheim Investigational Site 374, Tokushima Tokushima
  - Boehringer Ingelheim Investigational Site 375, Tokushima Tokushima
  - Boehringer Ingelheim Investigational Site 6, Tomakomai Hokkaido
  - Boehringer Ingelheim Investigational Site 380, Toon Ehime
  - Boehringer Ingelheim Investigational Site 71, Toride Ibaraki
  - Boehringer Ingelheim Investigational Site 220, Toyama Toyama
  - Boehringer Ingelheim Investigational Site 221, Toyama Toyama
  - Boehringer Ingelheim Investigational Site 263, Toyohashi Aichi
  - Boehringer Ingelheim Investigational Site 308, Toyonaka Osaka
  - Boehringer Ingelheim Investigational Site 273, Toyota Aichi
  - Boehringer Ingelheim Investigational Site 279, Tsu Mie
  - Boehringer Ingelheim Investigational Site 66, Tsuchiura Ibaraki
  - Boehringer Ingelheim Investigational Site 67, Tsuchiura Ibaraki
  - Boehringer Ingelheim Investigational Site 68, Tsuchiura Ibaraki
  - Boehringer Ingelheim Investigational Site 69, Tsukuba Ibaraki
  - Boehringer Ingelheim Investigational Site 72, Tsukuba Ibaraki
  - Boehringer Ingelheim Investigational Site 55, Tsuruoka Yamagata
  - Boehringer Ingelheim Investigational Site 354, Tsuyama Okayama
  - Boehringer Ingelheim Investigational Site 370, Ube Yamaguchi
  - Boehringer Ingelheim Investigational Site 240, Ueda Nagano
  - Boehringer Ingelheim Investigational Site 290, Uji Kyoto
  - Boehringer Ingelheim Investigational Site 431, Urasoe Okinawa
  - Boehringer Ingelheim Investigational Site 404, Ureshino Saga
  - Boehringer Ingelheim Investigational Site 81, Utsunomiya Tochigi
  - Boehringer Ingelheim Investigational Site 82, Utsunomiya Tochigi
  - Boehringer Ingelheim Investigational Site 344, Wakayama Wakayama
  - Boehringer Ingelheim Investigational Site 412, Yamaga Kumamoto
  - Boehringer Ingelheim Investigational Site 49, Yamagata Yamagata
  - Boehringer Ingelheim Investigational Site 50, Yamagata Yamagata
  - Boehringer Ingelheim Investigational Site 51, Yamagata Yamagata
  - Boehringer Ingelheim Investigational Site 52, Yamagata Yamagata
  - Boehringer Ingelheim Investigational Site 197, Yamato Kanagawa
  - Boehringer Ingelheim Investigational Site 401, Yanagawa Fukuoka
  - Boehringer Ingelheim Investigational Site 319, Yao Osaka
  - Boehringer Ingelheim Investigational Site 320, Yao Osaka
  - Boehringer Ingelheim Investigational Site 276, Yokkaichi Mie
  - Boehringer Ingelheim Investigational Site 277, Yokkaichi Mie
  - Boehringer Ingelheim Investigational Site 187, Yokohama Kanagawa
  - Boehringer Ingelheim Investigational Site 188, Yokohama Kanagawa
  - Boehringer Ingelheim Investigational Site 189, Yokohama Kanagawa
  - Boehringer Ingelheim Investigational Site 190, Yokohama Kanagawa
  - Boehringer Ingelheim Investigational Site 191, Yokohama Kanagawa
  - Boehringer Ingelheim Investigational Site 194, Yokohama Kanagawa
  - Boehringer Ingelheim Investigational Site 195, Yokohama Kanagawa
  - Boehringer Ingelheim Investigational Site 196, Yokohama Kanagawa
  - Boehringer Ingelheim Investigational Site 199, Yokohama Kanagawa
  - Boehringer Ingelheim Investigational Site 200, Yokohama Kanagawa
  - Boehringer Ingelheim Investigational Site 192, Yokosuka Kanagawa
  - Boehringer Ingelheim Investigational Site 193, Yokosuka Kanagawa
  - Boehringer Ingelheim Investigational Site 345, Yonago Tottori
  - Boehringer Ingelheim Investigational Site 229, Yoshida Fukui
  - Boehringer Ingelheim Investigational Site 230, Yoshida Fukui
  - Boehringer Ingelheim Investigational Site 400, Yukuhashi Fukuoka

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Case Report Form (CRF) collected for 1605 patients, 1602 added in safety set. 1 patient excluded due to out of contract period, 1 due to no treatment (with GIOTRIF) and 1 patient received (GIOTRIF) treatment before registration (total 3 patients excluded from the safety set). Participant flow is based on safety set.
Pre-assignment Details: This was a non-interventional, prospective, observational, single arm study based on new data collection.
Groups:
- Afatinib Dimaleate: The patients were administered single daily dose of Afatinib dimaleate tablet (GIOTRIF® Tablets), starting at 40 milligram (mg) orally up to a period of 52 weeks. The dosage might be adjusted according to the patient's tolerability, with a maximum daily dose of 50 mg.
Period: Overall Study
Arm/Group | Afatinib Dimaleate
Started | 1602 (Patients received treatment of GIOTRIF® Tablets)
Completed | 377 (Completed is defined as 52 weeks follow-up after starting administration of GIOTRIF® tablets.)
Not Completed | 1225
Not completed — Progressive disease | 751
Not completed — Adverse Event | 341
Not completed — Lost to Follow-up | 7
Not completed — Relocation | 32
Not completed — Other | 63
Not completed — Progressive disease/Adverse Event (AE) | 22
Not completed — Progressive disease/relocation | 1
Not completed — Progressive disease/other | 2
Not completed — AE/lost to follow-up | 1
Not completed — AE/other | 1
Not completed — Progressive disease/AE/other | 1
Not completed — Missing | 3

BASELINE CHARACTERISTICS:
Population: Safety Set: This analysis set included all patients who had received treatment of GIOTRIF® tablets except those who were found not following registration rules, invalid contract or previous treatment experience with GIOTRIF® tablets.
Arm/Group | Afatinib Dimaleate
Number analyzed (Participants) | 1602
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 947
  Male | 655

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Drug Reactions (ADRs)
Description: This outcome measure presents incidence of adverse drug reactions (ADRs). An ADR was defined as an AE if either the investigator or the sponsor (or both) assessed the causal relationship to GIOTRIF® Tablets either as "Yes", "Probably yes" or "Can't be denied".
  The number of patients with Adverse Drug Reactions (ADRs): "Malignant progression" reported as ADRs were included.
Time Frame: From first drug administration until 28 days after the last drug administration, up to 52 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Afatinib Dimaleate
Number analyzed (Participants) | 1602
Percentage of Participants | 95.19

2. Secondary Outcome: Objective Overall Response Based on Physician's Assessment [According to RECIST Version 1.1]
Description: Objective overall response based on investigator's assessment (according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for target lesions and assessed by MRI: complete response (CR) is the disappearance of all target lesions, a partial response (PR) is defined as at least a 30% decrease in the sum of the target lesion and stable disease (SD) is defined as fitting the criteria neither for progressive disease (PD) nor a PR. The population included the Tyrosine Kinase Inhibitor [TKI]-naïve patients and the TKI pre-treated patients.
  Overall response was calculated with 95% Clopper-Pearson confidence interval.
  OR = (CR+PR)/(CR+PR+SD+PD+Unknown)*100.
Time Frame: 52 weeks.
Population: Efficacy Set: This analysis set was a subset of the safety set, which included all patients in the safety set except those who had no available tumour assessment and/or who did not suffer from Epidermal Growth Factor Receptor (EGFR) mutation-positive inoperable or recurrent Non-Small Cell Lung Cancer (NSCLC).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib Dimaleate
Number analyzed (Participants) | 1602
Percentage of participants | 40.07 [37.66 to 42.52]

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after the last drug administration, up to 52 weeks.
Description: The number of participants presented in "Serious Adverse Events" and "Other Adverse Events" includes subjects with progressive disease.
Arm/Group | Afatinib Dimaleate
Serious Adverse Events (participants affected / at risk) | 1129/1602
Other Adverse Events (participants affected / at risk) | 1432/1602
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib Dimaleate (N=1602)
Anaemia (Blood and lymphatic system disorders) | 9
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Pericardial effusion (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Arrhythmia supraventricular (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Adrenal mass (Endocrine disorders) | 1
Retinal detachment (Eye disorders) | 2
Diplopia (Eye disorders) | 1
Iridocyclitis (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 117
Stomatitis (Gastrointestinal disorders) | 26
Vomiting (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 14
Enterocolitis (Gastrointestinal disorders) | 5
Ileus (Gastrointestinal disorders) | 5
Ileus paralytic (Gastrointestinal disorders) | 3
Melaena (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 1
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1
Oral disorder (Gastrointestinal disorders) | 1
Malaise (General disorders) | 12
Pyrexia (General disorders) | 9
General physical health deterioration (General disorders) | 3
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 2
Asthenia (General disorders) | 1
Feeling abnormal (General disorders) | 1
Gait disturbance (General disorders) | 1
Performance status decreased (General disorders) | 1
Inflammation (General disorders) | 1
Disuse syndrome (General disorders) | 1
Liver disorder (Hepatobiliary disorders) | 4
Hepatic failure (Hepatobiliary disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 3
Jaundice cholestatic (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Paronychia (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 6
Meningitis (Infections and infestations) | 4
Pneumonia bacterial (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 3
Lung infection (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Encephalitis (Infections and infestations) | 1
Gastroenteritis staphylococcal (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Pneumonia cryptococcal (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 6
Amylase increased (Investigations) | 3
Blood urea increased (Investigations) | 2
Carcinoembryonic antigen increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Lipase increased (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Transaminases increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 50
Dehydration (Metabolism and nutrition disorders) | 35
Feeding disorder (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 2
Hypophagia (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 813
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 27
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung infiltration malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 5
Depressed level of consciousness (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 3
Altered state of consciousness (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 2
Cerebellar haemorrhage (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
IIIrd nerve paralysis (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Monoparesis (Nervous system disorders) | 1
Monoplegia (Nervous system disorders) | 1
Paralysis (Nervous system disorders) | 1
Temporal lobe epilepsy (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Eating disorder (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Adjustment disorder (Psychiatric disorders) | 1
Renal impairment (Renal and urinary disorders) | 6
Acute kidney injury (Renal and urinary disorders) | 6
Renal disorder (Renal and urinary disorders) | 3
Prerenal failure (Renal and urinary disorders) | 3
Renal failure (Renal and urinary disorders) | 1
Renal infarct (Renal and urinary disorders) | 1
Ureteric rupture (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 60
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 9
Acne (Skin and subcutaneous tissue disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Aortic dissection (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Trousseau's syndrome (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib Dimaleate (N=1602)
Diarrhoea (Gastrointestinal disorders) | 1173
Stomatitis (Gastrointestinal disorders) | 473
Nausea (Gastrointestinal disorders) | 116
Paronychia (Infections and infestations) | 533
Decreased appetite (Metabolism and nutrition disorders) | 180
Rash (Skin and subcutaneous tissue disorders) | 644
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 183
Acne (Skin and subcutaneous tissue disorders) | 126
Dry skin (Skin and subcutaneous tissue disorders) | 83

LIMITATIONS AND CAVEATS:
The general scientific objective of this non-interventional study was to obtain an estimate of occurrence of AEs in the population under study. This study did not include a comparator, hindering the ability to this real world data into perspective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes